CLINICAL TRIAL: NCT06534619
Title: Additional Effects of Joint Mobilization in Addition to Rocabado Exercises on Alleviating Trismus Following Third Molar Extraction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/18
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Trismus
MeSH Terms: conditions — Trismus | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trail, having two groups. One group will receive Maitland joint mobilization along with rocabado exercises and the second will receive rocabado exercises only. Both groups will be recruited concurrently.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maitland joint mobilization + Rocabdo exercises (Experimental): Therapeutic ultrasound: pulse mode - 1:4, frequency 3 MHz, intensity- 0.8 watt/cm2 for about 3-4 Minutes.
  Mobilizations will be performed in Grade 1 initially and then progressed to Grade 2 and 3.
  Techniques used are anterior, lateral and inferior glides Frequency: 3-4 times in 1 week . 4 sessions in total.
  Interventions: Procedure: Electrotherapy; Procedure: Rocabado exercises; Procedure: Maitland oscillatory mobilizations
- Rocabado exercises (Experimental): Participants of this Group will receive the conventional physical therapy along with 6 Rocabado exercises.6 reps each Therapeutic ultrasound: pulse mode - 1:4, frequency 3 MHz, intensity- 0.8 watt/cm2 for about 3-4 Minutes.
  Frequency: 3-4 times in 1 week . 4 sessions in total.
  Interventions: Procedure: Electrotherapy; Procedure: Rocabado exercises

INTERVENTIONS:
Procedure: Electrotherapy — Therapeutic ultrasound: pulse mode - 1:4, frequency 3 MHz, intensity- 0.8 watt/cm2 for about 3-4 minutes.
Procedure: Rocabado exercises — 6 Rocabado exercises 6 Reps each.
Procedure: Maitland oscillatory mobilizations — Mobilizations will be performed in Grade 1 initially and then progressed to Grade 2 and 3.
  Techniques used are anterior, lateral and inferior glides
  Arms: Maitland joint mobilization + Rocabdo exercises

SUMMARY:
Without appropriate early intervention, prolonged trismus can lead to lasting complications like reduced jaw mobility or temporomandibular joint disorders.Therefore joint mobilization will impact on trismus, that will offer valuable insights into how these interventions will affect inflammation, muscle function and overall healing process within TMJ besides rocabado exercises that involves a series of movements and stretches targeting the muscles and joints involved in chewing,swallowing and speaking and minimizing muscle tension and opening the mouth, preventing further deterioration of jaw function and improving overall quality of life of individuals. If found effective, this will be added to the literature for the treatment of trismus after third molar extraction.

ELIGIBILITY:
Inclusion Criteria:

* Referral or consultation from a dentist to confirm the diagnosis of trismus.
* Age 18-45 years
* Both genders (Male and Female)
* Maximal interincisal opening ≤ 35mm (Restricted jaw motion).
* Unilateral/Bilateral impacted lower third molars.
* 3 days Post mandibular Third molar extraction

Exclusion Criteria:

* Local Infection or bleeding post third molar extraction.
* Patients with Acute pericoronitis
* Patient undergoing chemotherapy and radiotherapy.
* Type I diabetes, renal failure and chronic liver disease were excluded as immunocompromised state.
* Pregnant or lactating women.
* Cyst or tumor associated with impacted tooth

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 1 week
  pain will be measured using Numeric pain rating scale
Range of motion | 1 week
  A Vernier caliper will be used to measure maximal incisal opening (MIO) ≤ 35 mm (ROM)
Functional Performance | 1 week
  Gothenburg Trismus Questionnaire will be used for assessing functional performance or trismus-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan